CLINICAL TRIAL: NCT05294419
Title: The Healthcare Evaluation of Absolute Risk Testing Study: A Multi-centre, Single Arm, Pragmatic Study in Primary Care Setting
Brief Title: The Healthcare Evaluation of Absolute Risk Testing Study
Acronym: HEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genomics PLC (Industry)
Collaborators: NHS North of England Commissioning Support (NECS) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GEN2020-02
Record Dates: First submitted 2021-12-10; First posted 2022-03-24 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Per participant - cardiovascular integrated risk score (CVD-IRT) (Other): The CVD IRT device will generate a result based on the polygenic risk score derived from participant genomic and phenotypic information
  Interventions: Device: CVD Integrated Risk Test

INTERVENTIONS:
Device: CVD Integrated Risk Test — CVD IRT (Cardiovascular Integrated Risk Tool)

SUMMARY:
The aim of this study is to demonstrate the integration and use of cardiovascular disease (CVD) integrated risk tool (IRT) in an environment as close to real-world as possible.

This study will recruit participants of both biological sexes and any ancestry or background who require and are eligible for a CVD risk assessment as part of the NHS Health Check. Those aged 45-64 years are most likely to benefit from CVD IRT and will be included in the study, as they are more likely to be asymptomatic but also derive most benefit from preventative measures.

The study will be conducted in GP surgeries as the CVD IRT will have its greatest impact if incorporated into primary care practice for early identification of patients at highest risk.

This study is a device performance evaluation.

DETAILED DESCRIPTION:
The aim of this study is to demonstrate the integration and use of a cardiovascular disease (CVD) integrated risk tool (IRT) in an environment as close to real-world as possible.

In association with the routine healthchecks for CVD, the QRISK score will be integrated with the individuals polygenic risk score (from a blood sample) to produce the CVD IRT score, this score estimates the risk of CVD in the following 10years.

This study will recruit participants of both biological sexes and any ancestry or background who require and are eligible for a CVD risk assessment as part of the NHS Health Check. Those aged 45-64 years are most likely to benefit from CVD IRT and will be included in the study, as they are more likely to be asymptomatic but also derive most benefit from preventative measures.

The study will be conducted in GP surgeries as the CVD IRT will have its greatest impact if incorporated into primary care practice for early identification of patients at highest risk.

This study is a device performance evaluation. 1000 participants are expected to be enrolled. Of this, it is expected that 200 surveys will be completed and from those surveyed 20-30 interviewed. This would be considered an adequate determination of feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent and to comply with the study protocol
* Either male or female (biological sex)
* Aged 45-64 years (inclusive)
* Any ancestry or background
* Eligible for NHS Health Check using QRISK®2 assessment

Exclusion Criteria:

* Those excluded from NHS Health Checks;
* Currently prescribed and taking HMG-CoA reductase inhibitors (lipid-lowering preventive treatments or statins) for any indication.

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 862 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A Fuat, Prof, Principal Investigator — Carmel Medical Practice
Locations (1):
- Carmel Medical Practice, Darlington, Co Durham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled 836 participants from 12 sites, of which 832 participated in the analyses by providing blood samples and answering questionnaires. Of these participants 21 took part in the telephone interview. 23 HCPs took part in the final questionnaire, 12 HCPs took part in focus groups and 1 HCP completed an interview. Two PCCs took part in a focus group and 1 PCC completed an interview.
Groups:
- Participants Receiving CVD-IRT: Enrolled participants who elected to receive a CVD-IRT (Integrated Risk Tool reporting 10-year risk of CVD based on both QRISK2 and a PRS for CVD) as part of this study
- Healthcare Professionals (HCPs): HCPs who delivered CVD-IRT information to participants as part of this study
- Primary Care Commissioners (PCCs): PCCs who took part in this study (via focus group or interview)
Period: Overall Study
Arm/Group | Participants Receiving CVD-IRT | Healthcare Professionals (HCPs) | Primary Care Commissioners (PCCs)
Started | 836 | 23 | 3
Completed | 824 | 23 | 3
Not Completed | 12 | 0 | 0
Not completed — Protocol Violation | 4 | 0 | 0
Not completed — Lost to Follow-up | 6 | 0 | 0
Not completed — Results voided after publishing | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline measurements were only recorded for the "Participants Receiving CVD-IRT" arm. Baseline measurements were not recorded for the "Healthcare professionals (HCPs)" and "Primary care commissioners (PCCs)" arms.
Arm/Group | Participants Receiving CVD-IRT
Number analyzed (Participants) | 836
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 518
  Male | 318
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 813
  Mixed Multiple | 4
  Asian/ Asian British | 11
  Black: Africa/ Black Caribbean/ Black british | 4
  Other | 2
  NA | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 836

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Count of Participants Who Were Successfully Returned a Result
Description: Count of non-withdrawn participants (in "Participants Receiving CVD-IRT" arm) who were successfully returned a CVD-IRT result
Time Frame: 1.3-8.9 months from baseline (study enrolment)
Population: 836 were enrolled, 4 participants either withdrew or did not provide a sample for analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CVD-IRT
Number analyzed (Participants) | 832
Participants | 832

2. Primary Outcome: HCP Perception: Count of HCPs Recommending Test (End-of-study Questionnaire)
Description: Count of healthcare professionals responding "likely" or "very likely" in 5-point Likert response scale ("very unlikely" / "unlikely" / "undecided" / "likely" / "very likely") to the question "Would you recommend the test to colleagues in other practices?'" in HCP end-of-study questionnaire.
Time Frame: End of study (8-10 months after start of study)
Population: HCPs who delivered CVD-IRT information to participants as part of this study
Measure: Count of Participants; unit: Participants
Arm/Group | Healthcare Professionals (HCPs)
Number analyzed (Participants) | 23
Participants | 17

3. Primary Outcome: HCP Perception: Count of Favourable Ease-of-use Responses (Post-results Questionnaire)
Description: Count of "Yes" responses to the statement "The CVD-IRT can be incorporated into routine primary care in a straightforward manner" in the HCP post-results questionnaire (separate questionnaire filled at the time each CVD-IRT result was returned to participants)
Time Frame: 1.3-8.9 months from baseline (study enrolment)
Population: HCPs who delivered CVD-IRT information to participants as part of this study. A separate questionnaire was filled in every time a CVD-IRT result was returned.
Measure: Count of Units; unit: CVD-IRT results returned
Units Other Than Participants: CVD-IRT results returned
Arm/Group | Healthcare Professionals (HCPs)
Number analyzed (Participants) | 23
Number analyzed (CVD-IRT results returned) | 824
CVD-IRT results returned | 747

4. Primary Outcome: Participant Satisfaction: Count of Participants Recommending Test in Post-results Questionnaire
Description: Count of participants responding "likely" or "very likely" in Likert 5-point response scale ("very unlikely" / "unlikely" / "undecided" / "likely" / "very likely") to the question "How likely would you be to recommend the use of this test to friends or family in similar situations?" in the questionnaire given to participants after receiving their CVD-IRT results
Time Frame: 1.3-10 months from baseline (study enrolment)
Population: 520 participants responded after they received their CVD-IRT result, through an on-line survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CVD-IRT
Number analyzed (Participants) | 520
Participants | 452

5. Primary Outcome: Participant Satisfaction: Count of Participants Who Found Test Useful in Post-results Questionnaire
Description: Count of participants responding "Yes" to the question "Did you personally find this test useful?" in the questionnaire given to participants after receiving their CVD-IRT results
Time Frame: 1.3-10 months from baseline (study enrolment)
Population: 520 participants responded after they received their CVD-IRT result, through an on-line survey
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CVD-IRT
Number analyzed (Participants) | 520
Participants | 514

6. Primary Outcome: Participant Satisfaction: Count of Participants Who Found Test Easy to Understand in Post-results Questionnaire
Description: Count of participants responding "Yes" to the question "Were the results easy to understand?" in the questionnaire given to participants after receiving their CVD-IRT results
Time Frame: 1.3-10 months from baseline (study enrolment)
Population: 520 participants responded after they received their CVD-IRT result, through an on-line survey
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CVD-IRT
Number analyzed (Participants) | 520
Participants | 492

7. Primary Outcome: Feasibility: Result Return Time
Description: Time (in days) between study enrolment and receiving a CVD-IRT result (for participants in "Participants Receiving CVD-IRT" arm)
Time Frame: 1.3-8.9 months from baseline (study enrolment)
Population: 836 were enrolled, 4 participants either withdrew or did not provide a sample for analysis
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Participants Receiving CVD-IRT
Number analyzed (Participants) | 832
days | 60 [55 to 66]

8. Secondary Outcome: Risk Reclassification Counts
Description: Count of participants (in the "Participants Receiving CVD-IRT" arm) up-classified by the CVD-IRT (CVD-IRT≥10%, QRISK®2<10%) / down-classified by the CVD-IRT (CVD-IRT<10%, QRISK®2≥10%) / remained high risk (CVD-IRT≥10%, QRISK®2≥10%) / remained low risk (CVD-IRT<10%, QRISK®2<10%).
Time Frame: 1.3-8.9 months from baseline (study enrolment)
Population: 836 were enrolled, 4 participants either withdrew or did not provide a sample for analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CVD-IRT
Number analyzed (Participants) | 832
Participants
  Up-classified to high risk (CVD-IRT≥10%, QRISK®2<10%) | 43
  Down-classified to low risk (CVD-IRT<10%, QRISK®2≥10%) | 43
  Remained high risk for both CVD-IRT and QRISK®2 (≥10%) | 118
  Remained low risk for both CVD-IRT and QRISK®2 (<10%) | 628

9. Secondary Outcome: CVD-IRT Mean Value
Description: Mean risk score value (in the "Participants Receiving CVD-IRT" arm) of the CVD-IRT score
Time Frame: 1.3-8.9 months from baseline (study enrolment)
Population: 836 were enrolled, 4 participants either withdrew or did not provide a sample for analysis
Measure: Mean (Full Range); unit: percentage risk
Arm/Group | Participants Receiving CVD-IRT
Number analyzed (Participants) | 832
percentage risk | 6.6 [0.3 to 37.8]

10. Secondary Outcome: HCP Impact: Count of Changed Management Decisions (Post-results Questionnaire)
Description: Count of "Yes" responses to the statement "If the participant's CVD IRT score was greater than the participant's QRISK2 score, did this influence your management decision?" in the HCP post-results questionnaire (separate questionnaire filled at the time each CVD-IRT result was returned to participants) - responses were only recorded if CVD-IRT> QRISK2
Time Frame: 1.3-8.9 months from baseline (study enrolment)
Population: HCPs who delivered CVD-IRT information to participants as part of this study. A separate questionnaire was filled in every time a CVD-IRT result was returned. This question was only posed if CVD-IRT<QRISK2, a condition which was met for 388 results.
Measure: Count of Units; unit: CVD-IRT>QRISK2 results
Units Other Than Participants: CVD-IRT>QRISK2 results
Arm/Group | Healthcare Professionals (HCPs)
Number analyzed (Participants) | 23
Number analyzed (CVD-IRT>QRISK2 results) | 388
CVD-IRT>QRISK2 results | 108

11. Secondary Outcome: Participant Perception: Count of Participants Who Agreed Genetics is Important in Post-results Questionnaire
Description: Count of participants responding "agree" or "strongly agree" in Likert 5-point response scale ("strongly disagree" / "disagree" / "neither agree not disagree" / "agree" / "strongly agree") to the statement "When it comes to the risk of developing heart disease, genetics are as important to measure as factors such as blood pressure" in the questionnaire given to participants after receiving their CVD-IRT results
Time Frame: 1.3-10 months from baseline (study enrolment)
Population: 520 participants responded after they received their CVD-IRT result, through an on-line survey
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CVD-IRT
Number analyzed (Participants) | 520
Participants | 443

12. Secondary Outcome: Correlation in Saliva-derived and Blood-derived CVD-IRT Scores
Description: Some participants donated a saliva sample in addition to the blood sample (the primary DNA collection method used in this study). At the end of the study, CVD-IRT scores were also calculated from the saliva samples, and these were correlated against the blood-derived CVD-IRT scores
Time Frame: End of study (8-10 months after start of study)
Population: 91 participants donated a saliva sample in addition to the blood sample which was the primary DNA collection method in this study
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | Participants Receiving CVD-IRT
Number analyzed (Participants) | 91
Pearson correlation coefficient | 0.999

13. Secondary Outcome: Safety: Count of Participants Reporting Device Related Adverse Events or Deficiencies
Description: Safety: Count of participants reporting device related adverse events or deficiencies
Time Frame: From start of study to end of study (10 months after start of study)
Population: 836 were enrolled, 4 participants either withdrew or did not provide a sample for analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CVD-IRT
Number analyzed (Participants) | 836
Participants | 0

14. Secondary Outcome: QRISK®2 Mean Value
Description: Mean risk score value (in the "Participants Receiving CVD-IRT" arm) of the QRISK®2 score
Time Frame: Within 6 months of study enrolment
Population: 836 were enrolled, 4 participants either withdrew or did not provide a sample for analysis
Measure: Mean (Full Range); unit: percentage risk
Arm/Group | Participants Receiving CVD-IRT
Number analyzed (Participants) | 832
percentage risk | 6.4 [0.6 to 35.5]

ADVERSE EVENTS:
Time Frame: From start of study to end of study (10 months after start of study)
Description: The adverse event and device deficiency definitions were aligned to those in the international standard ISO 20916: 2019 for in vitro diagnostic medical devices. HCPs and PCCs were not monitored/assessed for Adverse Events per-protocol.
Arm/Group | Participants Receiving CVD-IRT
All-Cause Mortality (participants affected / at risk) | 0/836
Serious Adverse Events (participants affected / at risk) | 0/836
Other Adverse Events (participants affected / at risk) | 0/836

LIMITATIONS AND CAVEATS:
Planned rather than conducted changes in management practices were evaluated. Per protocol, HCPs delivered standard of care if the IRT produced a lower 10-year risk than QRISK. As a consequence, we did not assess potential changes in management when the inclusion of the PRS reduced overall risk. This study did not include an independent control group, so references to association only, rather than causation, regarding clinical decision making may be stated here.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT05294419/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT05294419/SAP_001.pdf